CLINICAL TRIAL: NCT04587388
Title: Towards Personalized Medicine for Refractory/Relapsed Follicular Lymphoma Patients: the Cantera/Lupiae Registry
Acronym: LUPIAE
Status: Recruiting | Type: Observational
Sponsor: European Hematology Association - Lymphoma Group (Other)
Collaborators: Associazione Angela Serra per la ricerca sul cancro (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor
Other Study IDs: W18_431
Record Dates: First submitted 2020-10-08; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Follicular Lymphoma; Relapsed/Refractory Follicular Lymphoma
Keywords: follicular lymphoma; relapsed/refractory disease; survival
MeSH Terms: conditions — Lymphoma, Follicular; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Histological block or slides for confirming the diagnosis. This analysis will be conducted retrospectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The optimal treatment strategy in patients with early progressive disease is not well known. In recent years, novel insights into the biology of Follicular Lymphoma (FL), and especially the role of the microenvironment, have resulted in the development of multiple novel treatment modalities. These new agents may ultimately improve the outlook for patients with FL with an unfavorable course, but for the development of the optimal therapeutic strategy, knowledge on the clinical and biological determinants of early refractory FL is needed.

DETAILED DESCRIPTION:
Patients with histologically confirmed follicular lymphoma are registered in the study at the time of the first event after first line treatment. An event is defined as refractory/relapsed disease documented by biopsy, imaging, or clinical evaluation. Registration is based on the locally established histological diagnosis, with exclusion of cases diagnosed on fine needle aspiration cytology, while tru-cut core-needle biopsies are permitted in the study. Registration will be done on-line on a key restricted accessible web-database: the Investigator must complete the on-line registration form after obtaining informed consent dated and signed by the patient.

Investigators are requested to register consecutive cases diagnosed at each participating Institution (all patients satisfying Inclusion criteria without any further selection). A patient number (Patient ID) will be assigned strictly sequentially in ascending order as patient's eligibility is verified. In case a patient's eligibility is not confirmed and the patient is withdrawn from the study, the patient number will not be reused. The assigned number will be used as the identification code for the subject.

Every registered case has to undergo histopathology review by a panel of experts. The reference pathologist will collect and review the pathology material sent by the participating centers, without knowledge of the clinical outcome of the patient. Both material obtained at diagnosis, and at relapse will be reviewed. Classification will be performed according to the World Health Organization recently published.

ELIGIBILITY:
Inclusion Criteria:

* Patients with initial diagnosis of follicular lymphoma, refractory/relapsed/transformed after first line therapy;
* All stages at the time of relapse;
* Histological grade 1-3a at the time of initial diagnosis;
* Age over 18 years;
* Availability of clinical data, including baseline information, comorbidities, data on disease localization, laboratory parameters at staging, features of treatment adopted and assurance of follow-up updating as requested
* Diagnostic material available for review;
* Written informed consent.

Exclusion Criteria:

• Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with initial diagnosis of follicular lymphoma, refractory/relapsed/transformed after first line therapy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-05-22 (Actual); Primary Completion 2023-05-22 (Estimated); Study Completion 2026-05-22 (Estimated)

PRIMARY OUTCOMES:
Rate of Progression of disease within 24 months from start of second line treatment (second POD24) | 24 months
  Second POD24 is defined as the rate of progression of disease at 24 months after the second line treatment.

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 and 5 years
  Overall Survival is measured from the date of diagnosis until death from any cause.
Progression-free survival after second line therapy (second PFS) | 3 and 5 years
  Second PFS is measured from the date of study entry until the date of disease progression or death from any cause.
Complete response rate at 30 months (CR30) from start of second line treatment (second CR30) | 30 months
  Second CR30 is defined as the rate of complete remissions at 30 months from start of second line treatment.

CONTACTS AND LOCATIONS:
Locations (11):
- Klinički Bolnički Centar Split, Split, Croatia
- AOU Città della Salute e della Scienza di Torino, Torino, Italy
- Netherlands (2):
  - Academic Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen
- Instituto Português de Oncologia Francisco Gentil, Lisbon, Portugal
- Spain (5):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Hospital Jose Maria Morales Meseguer, Murcia
  - Hospital de Son Llàtzer, Palma
  - Hospital Universitario de Salamanca, Salamanca
- Kiev National Cancer Institute, Kiev, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
We plan to share with other involved researchers the minimum information on IPD for publication.
  It is responsibility of the Study Coordinators to publish the study results after the completion of the study. It will be ensured that the data from one center are not published before the publication of the whole study. All publications regarding the results of the study will be marked with the sentence "on behalf of the EHA-LyG/Cantera-Lupiae study group". Participating centers and sites will be mentioned according to their overall contribution to the study, while all members of the study group will be included as authors of the manuscripts for their active contribution on the study design and procedures. No publication can occur without agreement of the study sponsor. Study results will be submitted for publication in peer-reviewed journals and for presentation at appropriate scientific meetings and conferences.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Preliminary analysis results will be made available during the study. Final results will be made available 6-12 months after the end of the study.

REFERENCES:
- [Background] Zelenetz AD, Gordon LI, Wierda WG, Abramson JS, Advani RH, Andreadis CB, Bartlett N, Byrd JC, Czuczman MS, Fayad LE, Fisher RI, Glenn MJ, Harris NL, Hoppe RT, Horwitz SM, Kelsey CR, Kim YH, Krivacic S, LaCasce AS, Nademanee A, Porcu P, Press O, Rabinovitch R, Reddy N, Reid E, Saad AA, Sokol L, Swinnen LJ, Tsien C, Vose JM, Yahalom J, Zafar N, Dwyer M, Sundar H; National comprehensive cancer network. Non-Hodgkin's lymphomas, version 4.2014. J Natl Compr Canc Netw. 2014 Sep;12(9):1282-303. doi: 10.6004/jnccn.2014.0125. PMID 25190696
- [Background] Swerdlow SH, Campo E, Pileri SA, Harris NL, Stein H, Siebert R, Advani R, Ghielmini M, Salles GA, Zelenetz AD, Jaffe ES. The 2016 revision of the World Health Organization classification of lymphoid neoplasms. Blood. 2016 May 19;127(20):2375-90. doi: 10.1182/blood-2016-01-643569. Epub 2016 Mar 15. PMID 26980727
- [Background] Mounier M, Bossard N, Remontet L, Belot A, Minicozzi P, De Angelis R, Capocaccia R, Iwaz J, Monnereau A, Troussard X, Sant M, Maynadie M, Giorgi R; EUROCARE-5 Working Group; CENSUR Working Survival Group. Changes in dynamics of excess mortality rates and net survival after diagnosis of follicular lymphoma or diffuse large B-cell lymphoma: comparison between European population-based data (EUROCARE-5). Lancet Haematol. 2015 Nov;2(11):e481-91. doi: 10.1016/S2352-3026(15)00155-6. Epub 2015 Oct 23. PMID 26686258
- [Background] Luminari S, Cesaretti M, Rashid I, Mammi C, Montanini A, Barbolini E, Bellei M, Pennese E, Sirotti MA, Marcheselli L, Partesotti G, Bari A, Maiorana A, Bonacorsi G, Federico M. Incidence, clinical characteristics and survival of malignant lymphomas: a population-based study from a cancer registry in northern Italy. Hematol Oncol. 2007 Dec;25(4):189-97. doi: 10.1002/hon.826. PMID 17654762
- [Background] Leich E, Ott G, Rosenwald A. Pathology, pathogenesis and molecular genetics of follicular NHL. Best Pract Res Clin Haematol. 2011 Jun;24(2):95-109. doi: 10.1016/j.beha.2011.02.003. Epub 2011 Apr 7. PMID 21658611
- [Background] de Jong D. Molecular pathogenesis of follicular lymphoma: a cross talk of genetic and immunologic factors. J Clin Oncol. 2005 Sep 10;23(26):6358-63. doi: 10.1200/JCO.2005.26.856. PMID 16155020
- [Background] Kuppers R. Mechanisms of B-cell lymphoma pathogenesis. Nat Rev Cancer. 2005 Apr;5(4):251-62. doi: 10.1038/nrc1589. PMID 15803153
- [Background] Kridel R, Sehn LH, Gascoyne RD. Pathogenesis of follicular lymphoma. J Clin Invest. 2012 Oct;122(10):3424-31. doi: 10.1172/JCI63186. Epub 2012 Oct 1. PMID 23023713
- [Background] Lossos IS, Gascoyne RD. Transformation of follicular lymphoma. Best Pract Res Clin Haematol. 2011 Jun;24(2):147-63. doi: 10.1016/j.beha.2011.02.006. Epub 2011 May 6. PMID 21658615
- [Background] Rowley JD. Chromosome studies in the non-Hodgkin's lymphomas: the role of the 14;18 translocation. J Clin Oncol. 1988 May;6(5):919-25. doi: 10.1200/JCO.1988.6.5.919. PMID 3284977
- [Background] Okosun J, Bodor C, Wang J, Araf S, Yang CY, Pan C, Boller S, Cittaro D, Bozek M, Iqbal S, Matthews J, Wrench D, Marzec J, Tawana K, Popov N, O'Riain C, O'Shea D, Carlotti E, Davies A, Lawrie CH, Matolcsy A, Calaminici M, Norton A, Byers RJ, Mein C, Stupka E, Lister TA, Lenz G, Montoto S, Gribben JG, Fan Y, Grosschedl R, Chelala C, Fitzgibbon J. Integrated genomic analysis identifies recurrent mutations and evolution patterns driving the initiation and progression of follicular lymphoma. Nat Genet. 2014 Feb;46(2):176-181. doi: 10.1038/ng.2856. Epub 2013 Dec 22. PMID 24362818
- [Background] Tan D, Horning SJ, Hoppe RT, Levy R, Rosenberg SA, Sigal BM, Warnke RA, Natkunam Y, Han SS, Yuen A, Plevritis SK, Advani RH. Improvements in observed and relative survival in follicular grade 1-2 lymphoma during 4 decades: the Stanford University experience. Blood. 2013 Aug 8;122(6):981-7. doi: 10.1182/blood-2013-03-491514. Epub 2013 Jun 18. PMID 23777769
- [Background] Bastion Y, Sebban C, Berger F, Felman P, Salles G, Dumontet C, Bryon PA, Coiffier B. Incidence, predictive factors, and outcome of lymphoma transformation in follicular lymphoma patients. J Clin Oncol. 1997 Apr;15(4):1587-94. doi: 10.1200/JCO.1997.15.4.1587. PMID 9193357
- [Background] Solal-Celigny P, Roy P, Colombat P, White J, Armitage JO, Arranz-Saez R, Au WY, Bellei M, Brice P, Caballero D, Coiffier B, Conde-Garcia E, Doyen C, Federico M, Fisher RI, Garcia-Conde JF, Guglielmi C, Hagenbeek A, Haioun C, LeBlanc M, Lister AT, Lopez-Guillermo A, McLaughlin P, Milpied N, Morel P, Mounier N, Proctor SJ, Rohatiner A, Smith P, Soubeyran P, Tilly H, Vitolo U, Zinzani PL, Zucca E, Montserrat E. Follicular lymphoma international prognostic index. Blood. 2004 Sep 1;104(5):1258-65. doi: 10.1182/blood-2003-12-4434. Epub 2004 May 4. PMID 15126323
- [Background] Federico M, Bellei M, Marcheselli L, Luminari S, Lopez-Guillermo A, Vitolo U, Pro B, Pileri S, Pulsoni A, Soubeyran P, Cortelazzo S, Martinelli G, Martelli M, Rigacci L, Arcaini L, Di Raimondo F, Merli F, Sabattini E, McLaughlin P, Solal-Celigny P. Follicular lymphoma international prognostic index 2: a new prognostic index for follicular lymphoma developed by the international follicular lymphoma prognostic factor project. J Clin Oncol. 2009 Sep 20;27(27):4555-62. doi: 10.1200/JCO.2008.21.3991. Epub 2009 Aug 3. PMID 19652063
- [Background] Murakami S, Kato H, Higuchi Y, Yamamoto K, Yamamoto H, Saito T, Taji H, Yatabe Y, Nakamura S, Kinoshita T. Prediction of high risk for death in patients with follicular lymphoma receiving rituximab plus cyclophosphamide, doxorubicin, vincristine, and prednisolone in first-line chemotherapy. Ann Hematol. 2016 Aug;95(8):1259-69. doi: 10.1007/s00277-016-2690-2. Epub 2016 May 25. PMID 27220639
- [Background] Tracy SI, Maurer MJ, Witzig TE, Drake MT, Ansell SM, Nowakowski GS, Thompson CA, Inwards DJ, Johnston PB, Micallef IN, Allmer C, Macon WR, Weiner GJ, Slager SL, Habermann TM, Link BK, Cerhan JR. Vitamin D insufficiency is associated with an increased risk of early clinical failure in follicular lymphoma. Blood Cancer J. 2017 Aug 25;7(8):e595. doi: 10.1038/bcj.2017.70. PMID 28841207
- [Background] Bachy E, Maurer MJ, Habermann TM, Gelas-Dore B, Maucort-Boulch D, Estell JA, Van den Neste E, Bouabdallah R, Gyan E, Feldman AL, Bargay J, Delmer A, Slager SL, Gomes da Silva M, Fitoussi O, Belada D, Maisonneuve H, Intragumtornchai T, Ansell SM, Lamy T, Dartigues P, Link BK, Seymour JF, Cerhan JR, Salles G. A simplified scoring system in de novo follicular lymphoma treated initially with immunochemotherapy. Blood. 2018 Jul 5;132(1):49-58. doi: 10.1182/blood-2017-11-816405. Epub 2018 Apr 17. PMID 29666118
- [Background] Huet S, Tesson B, Jais JP, Feldman AL, Magnano L, Thomas E, Traverse-Glehen A, Albaud B, Carrere M, Xerri L, Ansell SM, Baseggio L, Reyes C, Tarte K, Boyault S, Haioun C, Link BK, Feugier P, Lopez-Guillermo A, Tilly H, Brice P, Hayette S, Jardin F, Offner F, Sujobert P, Gentien D, Viari A, Campo E, Cerhan JR, Salles G. A gene-expression profiling score for prediction of outcome in patients with follicular lymphoma: a retrospective training and validation analysis in three international cohorts. Lancet Oncol. 2018 Apr;19(4):549-561. doi: 10.1016/S1470-2045(18)30102-5. Epub 2018 Feb 20. PMID 29475724
- [Background] Pastore A, Jurinovic V, Kridel R, Hoster E, Staiger AM, Szczepanowski M, Pott C, Kopp N, Murakami M, Horn H, Leich E, Moccia AA, Mottok A, Sunkavalli A, Van Hummelen P, Ducar M, Ennishi D, Shulha HP, Hother C, Connors JM, Sehn LH, Dreyling M, Neuberg D, Moller P, Feller AC, Hansmann ML, Stein H, Rosenwald A, Ott G, Klapper W, Unterhalt M, Hiddemann W, Gascoyne RD, Weinstock DM, Weigert O. Integration of gene mutations in risk prognostication for patients receiving first-line immunochemotherapy for follicular lymphoma: a retrospective analysis of a prospective clinical trial and validation in a population-based registry. Lancet Oncol. 2015 Sep;16(9):1111-1122. doi: 10.1016/S1470-2045(15)00169-2. Epub 2015 Aug 6. PMID 26256760
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753
- [Background] Dreyling M, Ghielmini M, Rule S, Salles G, Vitolo U, Ladetto M; ESMO Guidelines Committee. Newly diagnosed and relapsed follicular lymphoma: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2016 Sep;27(suppl 5):v83-v90. doi: 10.1093/annonc/mdw400. No abstract available. PMID 27664263
- [Background] Rummel MJ, Niederle N, Maschmeyer G, Banat GA, von Grunhagen U, Losem C, Kofahl-Krause D, Heil G, Welslau M, Balser C, Kaiser U, Weidmann E, Durk H, Ballo H, Stauch M, Roller F, Barth J, Hoelzer D, Hinke A, Brugger W; Study group indolent Lymphomas (StiL). Bendamustine plus rituximab versus CHOP plus rituximab as first-line treatment for patients with indolent and mantle-cell lymphomas: an open-label, multicentre, randomised, phase 3 non-inferiority trial. Lancet. 2013 Apr 6;381(9873):1203-10. doi: 10.1016/S0140-6736(12)61763-2. Epub 2013 Feb 20. PMID 23433739
- [Background] Federico M, Luminari S, Dondi A, Tucci A, Vitolo U, Rigacci L, Di Raimondo F, Carella AM, Pulsoni A, Merli F, Arcaini L, Angrilli F, Stelitano C, Gaidano G, Dell'olio M, Marcheselli L, Franco V, Galimberti S, Sacchi S, Brugiatelli M. R-CVP versus R-CHOP versus R-FM for the initial treatment of patients with advanced-stage follicular lymphoma: results of the FOLL05 trial conducted by the Fondazione Italiana Linfomi. J Clin Oncol. 2013 Apr 20;31(12):1506-13. doi: 10.1200/JCO.2012.45.0866. Epub 2013 Mar 25. PMID 23530110
- [Background] Federico M, Caballero Barrigon MD, Marcheselli L, Tarantino V, Manni M, Sarkozy C, Alonso-Alvarez S, Wondergem M, Cartron G, Lopez-Guillermo A, Issa D, Morschhauser F, Alcoceba M, Kimby E, Rusconi C, Chamuleau M, Holte H, Lockmer S, Montoto S, Gomes da Silva M, Aurer I, Zucca E, Paszkiewicz-Kozik E, Minoia C, Skrypets T, Blaker YN, Salles G, Coiffier B; Aristotle Consortium. Rituximab and the risk of transformation of follicular lymphoma: a retrospective pooled analysis. Lancet Haematol. 2018 Aug;5(8):e359-e367. doi: 10.1016/S2352-3026(18)30090-5. Epub 2018 Jul 4. PMID 30078408
- [Background] Sarkozy C, Trneny M, Xerri L, Wickham N, Feugier P, Leppa S, Brice P, Soubeyran P, Gomes Da Silva M, Mounier C, Offner F, Dupuis J, Caballero D, Canioni D, Paula M, Delarue R, Zachee P, Seymour J, Salles G, Tilly H. Risk Factors and Outcomes for Patients With Follicular Lymphoma Who Had Histologic Transformation After Response to First-Line Immunochemotherapy in the PRIMA Trial. J Clin Oncol. 2016 Aug 1;34(22):2575-82. doi: 10.1200/JCO.2015.65.7163. Epub 2016 Jun 13. PMID 27298402
- [Background] Trotman J, Luminari S, Boussetta S, Versari A, Dupuis J, Tychyj C, Marcheselli L, Berriolo-Riedinger A, Franceschetto A, Julian A, Ricard F, Guerra L, Haioun C, Biasoli I, Tilly H, Federico M, Salles G, Meignan M. Prognostic value of PET-CT after first-line therapy in patients with follicular lymphoma: a pooled analysis of central scan review in three multicentre studies. Lancet Haematol. 2014 Oct;1(1):e17-27. doi: 10.1016/S2352-3026(14)70008-0. Epub 2014 Sep 17. PMID 27030064
- [Background] Martinelli G, Schmitz SF, Utiger U, Cerny T, Hess U, Bassi S, Okkinga E, Stupp R, Stahel R, Heizmann M, Vorobiof D, Lohri A, Dietrich PY, Zucca E, Ghielmini M. Long-term follow-up of patients with follicular lymphoma receiving single-agent rituximab at two different schedules in trial SAKK 35/98. J Clin Oncol. 2010 Oct 10;28(29):4480-4. doi: 10.1200/JCO.2010.28.4786. Epub 2010 Aug 9. PMID 20697092
- [Background] Gopal AK, Kahl BS, de Vos S, Wagner-Johnston ND, Schuster SJ, Jurczak WJ, Flinn IW, Flowers CR, Martin P, Viardot A, Blum KA, Goy AH, Davies AJ, Zinzani PL, Dreyling M, Johnson D, Miller LL, Holes L, Li D, Dansey RD, Godfrey WR, Salles GA. PI3Kdelta inhibition by idelalisib in patients with relapsed indolent lymphoma. N Engl J Med. 2014 Mar 13;370(11):1008-18. doi: 10.1056/NEJMoa1314583. Epub 2014 Jan 22. PMID 24450858
- [Background] Montoto S, Corradini P, Dreyling M, Ghielmini M, Kimby E, Lopez-Guillermo A, Mackinnon S, Marcus RE, Salles G, Schouten HC, Sureda A, Dreger P. Indications for hematopoietic stem cell transplantation in patients with follicular lymphoma: a consensus project of the EBMT-Lymphoma Working Party. Haematologica. 2013 Jul;98(7):1014-21. doi: 10.3324/haematol.2013.084723. PMID 23813647
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krle A-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 Statement: defining standard protocol items for clinical trials. Rev Panam Salud Publica. 2015 Dec;38(6):506-14. PMID 27440100